CLINICAL TRIAL: NCT03913728
Title: Methotrexate Use Improvement in Rheumatoid Arthritis Using Biomarker Feedback: A Feasibility Trial
Brief Title: Methotrexate Use Improvement in Rheumatoid Arthritis Using Biomarker Feedback
Acronym: MIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr. James Bluett, Clinical Senior Lecturer, University of Manchester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS001485
Record Dates: First submitted 2019-03-28; First posted 2019-04-12 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Other clinical trial to study a novel intervention or randomised clinical trial to compare interventions in clinical practice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Outcome of blood test provided (Experimental): These patients are given the results of their drug level blood tests and treatment can be altered/ further advice can be provided as a result of this.
  Interventions: Other: Drug level blood tests
- Outcome of blood test not provided (No Intervention): The blood results for these people are not fed back to the patient or the clinical site.
- Patients have a telephone interview (Experimental): All patients are randomised for a second time; 20% (10) of them will have a semi-structured phone interview
  Interventions: Other: Telephone Interview
- No telephone interview (No Intervention): All patients are randomised for a second time; 80% won't have a phone call and this will be as per standard care.

INTERVENTIONS:
Other: Drug level blood tests — All information included previously.
  Arms: Outcome of blood test provided
Other: Telephone Interview — All information included previously.
  Arms: Patients have a telephone interview

SUMMARY:
The study is a prospective single-centre randomised controlled trial to examine the feasibility of a fully powered randomised controlled trial to examine if HPLC-SRM-MS guided intervention is superior to standard clinical care in improving clinical, behavioural and health-economy outcomes in RA patients prescribed MTX.

The trial will consist of 4 stages:

* Screening (~-2 weeks)
* Recruitment, consent, randomisation, data collection, examination and blood sampling - baseline visit 1 (time point 0)
* Intervention - telephone appointment (visit 2, intervention arm)
* Outcome - visit 3
* Process evaluation - visit 4

Prior to any trial specific procedures, the participant must have signed the informed consent form (ICF).

The trial will offer a small financial compensation for successfully recruited patients toward the costs of parking/refreshments/travel costs/inconvenience related to attending visits

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) affects up to 1% of the adult population. It is a condition that is treatable by medications. Methotrexate (MTX) is the first-line therapy for RA however, up to 60% of patients prescribed MTX still have active RA. This puts these patients at higher risk of joint damage compared to those whose RA is under control.

One important explanation for the poor control in those who receive treatment is that some patients, for many reasons, do not take their medications as recommended (non-adherence). Non-adherence is associated with increased costs to the NHS and reduced response to MTX.

The study will assess whether it is achievable to conduct a much larger study to explore whether a review of how well patients are coping with MTX can improve RA control. Understanding the reasons for poor RA control has the potential to improve the health and well-being of individual patients, avoid unnecessary tests and hospital appointments and save money in healthcare.

The trial will recruit 50 patients with RA who have been prescribed MTX for more than 2 years. 25 patients will be asked to donate blood samples and complete questionnaires, but their treatment will continue as standard. The blood tests will include patients MTX levels. The results of the test provide a direct measure of medication adherence. For the other 25 patients, the results of the blood tests will be fed back to them with tailored targeting of the main reason(s) for the deviation from the prescribed MTX. At the end of the study, the investigators will assess the feasibility of a randomised controlled trial of a biochemical screening of adherence guided intervention in patients with RA treated with MTX.

ELIGIBILITY:
Inclusion Criteria:

1. Prescribed oral MTX for ≥ two years
2. Clinical diagnosis of RA
3. Have a telephone
4. Male or female aged 18 years or above

Exclusion Criteria:

1. Patients with significant psychiatric illness as determined by the clinician
2. Patients unable to attend second appointment
3. Patients unable to provide informed consent
4. Patients with recent changes in the prescribed anti-rheumatic medications within 2 weeks of visit 1
5. Unable to speak English and complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Power for full randomized controlled trial | 3 months
  Change in proportion of people who adhere over 3 months
Patient opinion of HPLC-SRM-MS guided intervention using semi-structured interviewing | 1 year
Patient opinion of process of research, including outcome measures using semi-structured patient interviewing | 1 year
Number of patients correctly having intervention according to allocation | 1 year
Recruitment time | 1 year
  Length of time study needs to run for to recruit all participants
Number of patients invited to take part in the study and number of patients recruited | 1 year
Withdrawal rate | 1 year
Trial cost | 1 year

SECONDARY OUTCOMES:
Biochemical adherence | 1 year
  MTX quantified with HPLC-SRM-MS from serum.
DAS-28 at baseline and 3 months | 1 year
  The disease activity score-28 (DAS-28), range 2-10, higher values represent worse disease activity.
Quantity of patient encounters | 1 year
  Number of patient encounters with healthcare professionals per patient.

CONTACTS AND LOCATIONS:
Overall Officials: James Bluett, Principal Investigator — University of Manchester
Locations (1):
- Pennine MSK, Oldham, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No identifiable patient information will be shared with other researchers